CLINICAL TRIAL: NCT02583334
Title: Clinical Efficacy of Acupuncture in Patients With Fibromyalgia: A Multi-center, Randomized, Assessor and Participant-blinded, Controlled, and Parallel-design Clinical Trial
Brief Title: Acupuncture for Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH103-REC1-138
Record Dates: First submitted 2015-06-07; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Fibromyalgia
Keywords: acupuncture; fibromyalgia; rheumatism; clinical trial
MeSH Terms: conditions — Fibromyalgia; Rheumatic Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum Acupuncture (Experimental): After diagnosis by rheumatologist, participants will be randomized to receive verum acupuncture or sham acupuncture treatment. In the verum acupuncture group, participants will receive verum acupuncture (Device: 30# acupuncture needle) three times a week, for 4 weeks (12 treatment in total).
  Interventions: Device: Verum acupuncture (30# acupuncture needle)
- Sham Acupuncture (Sham Comparator): After diagnosis by rheumatologist, participants will be randomized to receive verum acupuncture or sham acupuncture treatment. In the sham acupuncture group, participants will receive sham acupuncture (Device: Streitberger device) three times a week, for 4 weeks (12 treatment in total).
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Verum acupuncture (30# acupuncture needle) — Acupuncture will be applied by inserting acupuncture needle into acupoints (LI4, LI11, LR3, ST36, SP6, GB34)
  Arms: Verum Acupuncture
Device: Sham acupuncture — Streitberger device will be applied by onto acupoints (LI4, LI11, LR3, ST36, SP6, GB34). The device will not really insert the blunt needle into skin but let the participants feel like real acupuncture (Lancet 1998; 352: 364-365.).
  Other Names: Streitberger device
  Arms: Sham Acupuncture

SUMMARY:
Fibromyalgia is the second most common autoimmune rheumatic diseases with clinical manifestations of widespread pain, fatigue and accompanied cognitive and emotional disturbances. It often associated with sleep disorders and headaches. The cardinal symptom of fibromyalgia is widespread pain. Clinical observations reveal that pain in patients with fibromyalgia could not simply improve by using analgesics only. Patients often use Chinese medicine or acupuncture to help them to ease the pain.

The aim of this study is to investigate the efficacy of acupuncture in patients with fibromyalgia. The study adapted a randomized, assessor- and participant-blinded, sham-controlled, and parallel-design approach to investigate whether acupuncture can improve the clinical symptoms and quality of life as well as the mechanism through laboratory biochemistric and image study.

DETAILED DESCRIPTION:
A total of 158 volunteers of patients with fibromyalgia will be recruited from the Chinese medicine or Western medicine clinics in China Medical University Hospital(Taichung and other affiliated branches). After diagnosis by rheumatologist, these patients will be randomized to receive verum acupuncture or sham acupuncture treatment, three times a week, for 4 weeks (12 treatment in total). Visual analogue scale will be done for every visit. Laboratory biochemistric analysis and other questionnaires including Visual Analogue Scale, Fibromyalgia Impact Questionnaire, SF-36 health survey, Pittsburgh Sleep Quality Index and Beck Depression Inventory-II will be completed at baseline, 2, 4 weeks after initiation of intervention (complete acupuncture treatment), 4 weeks after completion of acupuncture completion (8 weeks). PET image examination (optional; this item depends on patients' own will) and instrumental examinations including heart rate variability and traditional Chinese medicine four examinations will be given before and after intervention. We expect that the efficacy of verum acupuncture is superior to sham acupuncture in improving pain, fatigue, physical function and quality of life. The effectiveness of acupuncture can be detected by questionnaires. Moreover, we will further speculate the mechanism by analyzing laboratory and image data.

ELIGIBILITY:
Inclusion Criteria:

1. Participants met the diagnostic criteria (American College of Rheumatology, 2011) and were diagnosed fibromyalgia.
2. Persisted pain for more than 50 percent of time.
3. Adult volunteers of ages between 20~75 years old.
4. Male or female genders.
5. No allergy or contraindication to stainless needles.
6. Participants understood the aim and process of the trial, agreed to participate in trial as well as completed informed consent.

Exclusion Criteria:

1. More than 75 or less than 20 years old.
2. Had used opioid or narcotic analgesic drugs within one month before the beginning of trial.
3. Had used Pregabalin within 6 months.
4. Drug abuse.
5. Coagulation dysfunction or low platelet count in blood tests(platelet≤150000 / uL).
6. Other diagnosed rheumatoid comorbidities such as rheumatoid arthritis, systemic lupus erythema, inflammatory bowel disease, autoimmune thyroiditis.
7. Participating in other clinical trials.
8. Pregnancy or lactation.
9. Severe psychological or behavioral disorders such as schizophrenia.
10. Arrhythmia patients with pacer marker.
11. Severe diseases such as myocardial infarction, severe arrhythmia,cardiac arrest, chronic obstructive pulmonary disease, renal failure and cancers.
12. Limbs edema and severe skin lesions contraindicated to acupuncture.
13. Had Chinese medicine or acupuncture within two weeks prior to the beginning of trial.
14. Had not completed informed consent.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire | 0,2,4,8 week
  Changes from baseline to midpoint、end of intervention and 4 weeks after intervention completed

SECONDARY OUTCOMES:
SF-36 health survey | 0,2,4,8 week
  Changes from baseline to midpoint、end of intervention and 4 weeks after intervention completed
Pittsburgh Sleep Quality Index | 0,2,4,8 week
  Changes from baseline to midpoint、end of intervention and 4 weeks after intervention completed
Beck Depression Inventory-II | 0,2,4,8 week
  Changes from baseline to midpoint、end of intervention and 4 weeks after intervention completed
The Constitution in Chinese Medicine Questionnaire | 0,2,4,8 week
  Changes from baseline to midpoint、end of intervention and 4 weeks after intervention completed
Heart rate variability | 0,4 week
  Changes from baseline to the end of intervention
Laboratory examination: cytokines | 0,4 week
  Changes from baseline to the end of intervention
Hematogram | 0,4 week
  Changes from baseline to the end of intervention
FDG PET/CT scan | 0, 4-6week
  optional examination; changes from baseline to the 4-6week of intervention
Visual Analogue Scale | 0,2,4,8 week
  Changes from baseline to midpoint、end of intervention and 4 weeks after intervention completed
TCM four examinations | 0,4 week
  Changes from baseline to the end of intervention
Liver function test | 0,4 week
  Changes at baseline and end of intervention
Renal function test | 0,4 week
  Changes from baseline to the end of intervention
Widespread pain index | 0,2,4,8 week
  Changes from baseline to midpoint、end of intervention and 4 weeks after intervention completed
Symptom severity scale | 0,2,4,8 week
  Changes from baseline to midpoint、end of intervention and 4 weeks after intervention completed

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Rong Yen, M.D., Ph.D., Principal Investigator — China Medical University Hospital
Locations (2):
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - China Medical University Hospital-Taipei branch, Taipei